CLINICAL TRIAL: NCT00288743
Title: Adherence, Efficacy and Safety of an Insulin Protocol in the Critically Ill: A Prospective Observational Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2002/087
Record Dates: First submitted 2006-02-07; First posted 2006-02-08 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Critically Ill Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: to implement an insulin protocol with target blood glucose levels between 81-110 mg/dL.

SUMMARY:
There is a growing body of evidence in the literature regarding the adverse effects of hyperglycemia in critically ill patients. To target and maintain better blood glucose regulation we implemented an insulin protocol with target blood glucose levels between 81-110 mg/dL.

ELIGIBILITY:
Inclusion Criteria:

* Surgical or medical critically ill patients
* An expected ICU-stay of more than 72 hours
* Age > 16 years
* Need for insulin therapy
* Patients must have an arterial line

Exclusion Criteria:

* Patients who did not respond to the inclusion criteria
* Patients with diabetic ketoacidosis
* Cardiac surgical patients
* Patients transferred from other hospitals
* Other study enrollment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2002-09; Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
To evaluate compliance, efficacy and safety of an insulin protocol, with target glycemia between 81-110 mg/dL in critically ill patients

SECONDARY OUTCOMES:
To determine potential factors associated with blood glucose control

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Oeyen, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be